CLINICAL TRIAL: NCT04113499
Title: A Randomized Trial Comparing Direct Endoscopic Necrosectomy vs. Step-up Transluminal Endoscopic Interventions in Infected Necrotizing Pancreatitis (DESTIN)
Brief Title: Endoscopic Necrosectomy Versus Step-up Endoscopic Intervention
Acronym: DESTIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1438851
Record Dates: First submitted 2019-10-01; First posted 2019-10-02 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Pancreatic Necrosis; Necrosis Pancreas
Keywords: pancreatic necrosis; pancreatic necrotic collection; transenteric drainage; necrosectomy
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: During follow up, the coordinators that are contacting the subjects will be blinded to the randomization assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Direct Endoscopic Necrosectomy (Active Comparator): The subject will have endoscopic drainage and necrosectomy at the time of the index intervention.
  Interventions: Procedure: Direct Endoscopic Intervention
- Step-up Endoscopic Interventions (Active Comparator): The subject will only have endoscopic drainage of the pancreatic necrotic collection at the time of index intervention.
  Interventions: Procedure: Step-up Endoscopic Intervention

INTERVENTIONS:
Procedure: Direct Endoscopic Intervention — The necrotic collection is first identified using a linear echoendoscope. A Hot AXIOS stent is utilized in all patients for EUS-guided drainage of the necrotic collection. The necrotic material is sent for gram stain and culture with sensitivities.
  For endoscopic necrosectomy, in patients allocated to direct endoscopic necrosectomy group, endoscopic necrosectomy is performed during the same session as the index endoscopic drainage. It is performed using a therapeutic gastroscope and various accessories (see below for further details) for 90 to 120 minutes.
  Arms: Direct Endoscopic Necrosectomy
Procedure: Step-up Endoscopic Intervention — The necrotic collection is first identified using a linear echoendoscope. A Hot AXIOS stent is utilized in all patients for EUS-guided drainage of the necrotic collection. The necrotic material is sent for gram stain and culture with sensitivities.
  In patients allocated to the step-up endoscopic interventions group, endoscopic necrosectomy is not performed at the time of the index intervention, however it is performed when clinically indicated during the follow-up period (6 months from index intervention).
  Arms: Step-up Endoscopic Interventions

SUMMARY:
This trial is to compare clinical outcomes between patients undergoing immediate endoscopic necrosectomy compared to step-up endoscopic interventions in patients undergoing endoscopic therapy for infected necrotizing pancreatitis.

DETAILED DESCRIPTION:
Acute pancreatitis has an annual incidence of 13-45 cases per 100,000 persons and is one of the most common gastrointestinal disorders requiring hospitalization worldwide. It leads to over a quarter of a million hospital admissions annually in the United States, and inpatient costs exceeding 2.5 billion US dollars. Pancreatic necrosis occurs as a consequence of severe acute pancreatitis in approximately 20% of patients. It can mature into a contained necrotic collection, typically four weeks into the disease course. With intense conservative management, including nutritional and intensive care support when required, the collection may resolve without intervention. However, a persistent collection with pain, gastric outlet, intestinal or biliary obstruction, new-onset or persisting organ failure, persistent unwellness or infection is associated with a mortality of 15-20%, and requires necrosectomy and drainage. Without intervention, infected necrosis ultimately leads to death in nearly every patient.

Recently, there has been a shift away from surgical debridement (necrosectomy) towards minimally-invasive endoscopic methods in the treatment of necrotizing pancreatitis. Endoscopic management involves creation of a fistula between the enteric wall and necrotic collection under the guidance of endoscopic ultrasound [EUS] with subsequent placement of a stent to allow drainage of the necrotic material. Endoscopic transenteral drainage of necrotic collection is associated with favorable outcomes, with treatment success rates reported in the range of 45-70%. Endoscopic necrosectomy, with the additional technique of extraction of necrotic material under direct endoscopic visualization has increased rates of treatment success to greater than 80%.

However, there are currently scant data on the optimal timing of endoscopic necrosectomy. In a retrospective study, performing endoscopic necrosectomy at the time of the initial EUS-guided drainage of the necrotic collection was associated with a significantly lower number of necrosectomy sessions compared to performing endoscopic necrosectomy one week after drainage.

The aim of this randomized trial is to compare clinical outcomes between patients undergoing immediate endoscopic necrosectomy (direct endoscopic necrosectomy) compared to step-up endoscopic interventions in patients undergoing endoscopic therapy for infected necrotizing pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

1. The subject (or when applicable the subject's LAR) is capable of understanding and complying with protocol requirements
2. The subject (or when applicable the subject's LAR) is able to understand and willing to sign an informed consent form prior to the initiation of any study procedures
3. Males or females ≥ 18 years of age
4. Necrotic collection diagnosed on MRI or CT abdomen/pelvis (seen as a fluid collection in the setting of documented pancreatic necrosis that contains necrotic material and encased within a partial or complete wall)
5. Necrotic collection of any size with ≥ 33% of solid/necrotic component and any no. of loculations, located within the pancreatic/peri-pancreatic space
6. Necrotic collection visualized on EUS and amenable to EUS-guided drainage
7. Suspected/confirmed infected necrotic collection. Infected necrosis is defined by the presence of gas in the necrotic collection on cross-sectional imaging or positive culture of necrotic tissue obtained preprocedure or at first intervention. Infected necrosis is also suspected when sepsis is persistent or in the presence of ongoing clinical deterioration.
8. Documented history of acute pancreatitis Acute pancreatitis is diagnosed if 2 of the following 3 criteria are met

   1. Abdominal pain characteristic of acute pancreatitis
   2. Serum lipase/amylase ≥ x3 upper limit of normal
   3. Characteristic radiological findings of acute pancreatitis on CECT/MRI/US abdomen, such as homogeneous enhancement of pancreatic parenchyma, standing of peripancreatic fat
9. Able to undergo general anesthesia

Exclusion Criteria:

1. Females who are pregnant or lactating. Pregnancy for females of childbearing potential will be determined by routine preoperative urine or serum HCG testing.
2. Irreversible coagulopathy (INR >1.5, thrombocytopenia with platelet count <50,000/mL)
3. Has surgically altered gastrointestinal anatomy such as but not limited to Billroth II, Roux-en-Y, gastric bypass
4. Age < 18 years
5. Unable to obtain consent for the procedure from either the patient or LAR
6. Use of anticoagulants that cannot be discontinued for the procedure
7. Unable to tolerate general anesthesia
8. Necrotic collection that is not accessible for EUS-guided drainage
9. Percutaneous drainage of the necrotic collection is required or performed prior to EUS-guided drainage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-11-27 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-04-25 (Actual)

PRIMARY OUTCOMES:
Rate of treatment success | 6 months
  Treatment success is defined as the resolution of necrotic collection on CT scan in association with clinical resolution of symptoms at 6-month follow-up

SECONDARY OUTCOMES:
Rate of resolution of pre-intervention systemic inflammatory response syndrome | 72 hours post index procedure
  Assessment of preintervention systemic inflammatory response syndrome & their resolution and measured by yes/no.
Rate of resolution of at least 1 pre-intervention organ failure | 72 hours post index procedure
  Assessment of organ failure following the index procedure and their resolution and measured by yes/no.
Number of re-admissions | 6 months
  Assessing the total number of re-admissions following the index procedure.
Rate of technical success for EUS-guided cystogastrostomy | 24 hours
  Technical success for EUS-guided cystogastrostomy defined as completion of endoscopic necrosectomy session as planned without the occurrence of adverse events and measured by yes/no.
Rate of technical success for endoscopic necrosectomy | 6 months
  Technical success for endoscopic necrosectomy defined as any adverse event occurring as a result of necrotizing pancreatitis and measured by yes/no.
Rate of exocrine pancreatic insufficiency | 6 months
  Rate of exocrine pancreatic insufficiency defined as fecal elastase level < 200μg/g in patients not previously taking pancreatic enzyme supplements
Rate of new onset diabetes | 6 months
  Rate of new onset diabetes defined as new onset elevation in fasting plasma glucose ≥ 126 mg/dL, 2-hour plasma glucose ≥ 200 mg/dL after an oral glucose tolerance test or HbA1c ≥ 6.5%
Number of Procedure-related adverse events | 6 months
  Procedure-related adverse events defined as any adverse event occurring as a result of any endoscopic intervention. The subject will be asked to report and medical records will be reviewed for any adverse events related to the procedure.
Number of Disease-related adverse events | 6 months
  Disease-related adverse events, defined as any adverse event occurring as a result of necrotizing pancreatitis. The subject will be asked to report and medical records will be reviewed for any adverse events related to the procedure.
Post-procedure length of intensive care unit (ICU) stay | 6 months
  Measured in the number of days in the intensive care unit
Total length of hospital stay | 6 months
  Measured in the number of days in the hospital
Overall treatment costs | 6 months
  Overall treatment costs from admission until 6 months post index intervention. All relevant costs pertaining to treatment will be taken into consideration - procedure costs, inpatient hospital stay from date of procedure to discharge, readmissions, medications, materials, anesthesia, pharmacy and imaging studies.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Hasan, MD, Principal Investigator — AdventHealth
Locations (1):
- Center for Interventional Endoscopy, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yadav D, Lowenfels AB. The epidemiology of pancreatitis and pancreatic cancer. Gastroenterology. 2013 Jun;144(6):1252-61. doi: 10.1053/j.gastro.2013.01.068. PMID 23622135
- [Background] Peery AF, Dellon ES, Lund J, Crockett SD, McGowan CE, Bulsiewicz WJ, Gangarosa LM, Thiny MT, Stizenberg K, Morgan DR, Ringel Y, Kim HP, DiBonaventura MD, Carroll CF, Allen JK, Cook SF, Sandler RS, Kappelman MD, Shaheen NJ. Burden of gastrointestinal disease in the United States: 2012 update. Gastroenterology. 2012 Nov;143(5):1179-1187.e3. doi: 10.1053/j.gastro.2012.08.002. Epub 2012 Aug 8. PMID 22885331
- [Background] Beger HG, Rau B, Mayer J, Pralle U. Natural course of acute pancreatitis. World J Surg. 1997 Feb;21(2):130-5. doi: 10.1007/s002689900204. PMID 8995067
- [Background] Banks PA, Bollen TL, Dervenis C, Gooszen HG, Johnson CD, Sarr MG, Tsiotos GG, Vege SS; Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis--2012: revision of the Atlanta classification and definitions by international consensus. Gut. 2013 Jan;62(1):102-11. doi: 10.1136/gutjnl-2012-302779. Epub 2012 Oct 25. PMID 23100216
- [Background] van Brunschot S, Bakker OJ, Besselink MG, Bollen TL, Fockens P, Gooszen HG, van Santvoort HC; Dutch Pancreatitis Study Group. Treatment of necrotizing pancreatitis. Clin Gastroenterol Hepatol. 2012 Nov;10(11):1190-201. doi: 10.1016/j.cgh.2012.05.005. Epub 2012 May 18. PMID 22610008
- [Background] Bang JY, Arnoletti JP, Holt BA, Sutton B, Hasan MK, Navaneethan U, Feranec N, Wilcox CM, Tharian B, Hawes RH, Varadarajulu S. An Endoscopic Transluminal Approach, Compared With Minimally Invasive Surgery, Reduces Complications and Costs for Patients With Necrotizing Pancreatitis. Gastroenterology. 2019 Mar;156(4):1027-1040.e3. doi: 10.1053/j.gastro.2018.11.031. Epub 2018 Nov 16. PMID 30452918
- [Background] Gardner TB, Chahal P, Papachristou GI, Vege SS, Petersen BT, Gostout CJ, Topazian MD, Takahashi N, Sarr MG, Baron TH. A comparison of direct endoscopic necrosectomy with transmural endoscopic drainage for the treatment of walled-off pancreatic necrosis. Gastrointest Endosc. 2009 May;69(6):1085-94. doi: 10.1016/j.gie.2008.06.061. Epub 2009 Feb 24. PMID 19243764
- [Background] Varadarajulu S, Bang JY, Phadnis MA, Christein JD, Wilcox CM. Endoscopic transmural drainage of peripancreatic fluid collections: outcomes and predictors of treatment success in 211 consecutive patients. J Gastrointest Surg. 2011 Nov;15(11):2080-8. doi: 10.1007/s11605-011-1621-8. Epub 2011 Jul 23. PMID 21786063
- [Background] Yan L, Dargan A, Nieto J, Shariaha RZ, Binmoeller KF, Adler DG, DeSimone M, Berzin T, Swahney M, Draganov PV, Yang DJ, Diehl DL, Wang L, Ghulab A, Butt N, Siddiqui AA. Direct endoscopic necrosectomy at the time of transmural stent placement results in earlier resolution of complex walled-off pancreatic necrosis: Results from a large multicenter United States trial. Endosc Ultrasound. 2019 May-Jun;8(3):172-179. doi: 10.4103/eus.eus_108_17. PMID 29882517
- [Background] Bang JY, Navaneethan U, Hasan MK, Sutton B, Hawes R, Varadarajulu S. Non-superiority of lumen-apposing metal stents over plastic stents for drainage of walled-off necrosis in a randomised trial. Gut. 2019 Jul;68(7):1200-1209. doi: 10.1136/gutjnl-2017-315335. Epub 2018 Jun 1. PMID 29858393
- [Background] Bang JY, Hasan MK, Navaneethan U, Sutton B, Frandah W, Siddique S, Hawes RH, Varadarajulu S. Lumen-apposing metal stents for drainage of pancreatic fluid collections: When and for whom? Dig Endosc. 2017 Jan;29(1):83-90. doi: 10.1111/den.12681. Epub 2016 Jun 15. PMID 27199157
- [Derived] Bang JY, Lakhtakia S, Thakkar S, Buxbaum JL, Waxman I, Sutton B, Memon SF, Singh S, Basha J, Singh A, Navaneethan U, Hawes RH, Wilcox CM, Varadarajulu S; United States Pancreatic Disease Study Group. Upfront endoscopic necrosectomy or step-up endoscopic approach for infected necrotising pancreatitis (DESTIN): a single-blinded, multicentre, randomised trial. Lancet Gastroenterol Hepatol. 2024 Jan;9(1):22-33. doi: 10.1016/S2468-1253(23)00331-X. Epub 2023 Nov 18. PMID 37980922